CLINICAL TRIAL: NCT05675345
Title: Physiological Effects of Continuous Negative External Pressure for Acute Hypoxemic Respiratory Failure: A Pilot Crossover Trial
Brief Title: Physiological Effects of Continuous Negative External Pressure for Acute Hypoxemic Respiratory Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jeremy Beitler, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAAT7361
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: acute respiratory distress syndrome; noninvasive ventilation; mechanical ventilation; oxygen inhalation therapy; atelectasis; high-flow nasal cannula
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- HFNC only (Active Comparator)
  Interventions: Device: HFNC only
- HFNC + CNEP10 (Experimental)
  Interventions: Device: HFNC + CNEP10
- HFNC + CNEP20 (Experimental)
  Interventions: Device: HFNC + CNEP20
- HFNC + CNEP30 (Experimental)
  Interventions: Device: HFNC + CNEP30

INTERVENTIONS:
Device: HFNC only — HFNC for 45 minutes, with FiO2 titrated to SpO2 of 90-97%
  Arms: HFNC only
Device: HFNC + CNEP10 — HFNC with CNEP of 10 cmH2O for 45 minutes, with FiO2 titrated to SpO2 of 90-97%
  Arms: HFNC + CNEP10
Device: HFNC + CNEP20 — HFNC with CNEP of 20 cmH2O for 45 minutes, with FiO2 titrated to SpO2 of 90-97%
  Arms: HFNC + CNEP20
Device: HFNC + CNEP30 — HFNC with CNEP of 30 cmH2O for 45 minutes, with FiO2 titrated to SpO2 of 90-97%
  Arms: HFNC + CNEP30

SUMMARY:
This study is being conducted to evaluate if wearing a non-invasive breathing support device over the chest/abdomen improves markers of breathing in patients with lung injury requiring high-flow oxygen. The breathing support device consists of a plastic shell that sits over the chest and abdomen and connects to a vacuum that helps the chest expand with breathing. This breathing support is known as continuous negative external pressure (CNEP). Study findings will help determine if this breathing support device might be useful for patients with acute hypoxemic respiratory failure (AHRF).

DETAILED DESCRIPTION:
This study is a prospective randomized cross-over trial. Eligible, consenting participants will undergo 4 strategies of respiratory support: high-flow nasal cannula (HFNC) only, HFNC + continuous negative external pressure (CNEP) of 10 cmH2O, HFNC + CNEP of 20 cmH2O, HFNC + CNEP of 30 cmH2O. Throughout the study period, HFNC will be managed at a constant flow rate with fraction of inspired oxygen (FiO2) titrated to achieve goal oxygen saturation (SpO2) of 90-97%, measured via continuous pulse-oximetry. Each of the 4 strategies will be performed for 45 minutes per strategy, interspersed with a 15-minute washout period of HFNC only. Participants will be randomized to the sequence of strategies for respiratory support.

A summary of the sequence of trial procedures is as follows:

1. Perform baseline measures.
2. Wait 5-10 minutes for recovery.
3. Initiate first random treatment assignment for up to 45 minutes.
4. HFNC-only washout for 15 minutes
5. Initiate second random treatment assignment for up to 45 minutes.
6. HFNC-only washout for 15 minutes
7. Initiate third random treatment assignment for up to 45 minutes.
8. HFNC-only washout for 15 minutes
9. Initiate fourth random treatment assignment for up to 45 minutes.
10. Return to usual care (HFNC only)

If a participant does not tolerate a given level of CNEP, the patient will be returned to HFNC for 5 minutes and then given the option to attempt that CNEP level again. If the patient declines reattempt or does not tolerate that CNEP level on reattempt, the HFNC-only washout will be instituted for 15 minutes before proceeding to the next protocol step.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Acute hypoxemic respiratory failure
* Non-cardiogenic airspace opacities on chest radiograph or computed tomography (CT) scan
* High-flow nasal cannula (flow ≥ 30 LPM) initiated within last 96 hours (4 days)
* FiO2 ≥ 40%
* SpO2 ≥ 92%

Exclusion Criteria:

* Do-not-intubate order
* Anatomical factor predisposing to poor fit of cuirass (e.g. severe kyphosis or scoliosis)
* Use of cuirass precluded, e.g. due to:

  * Clinically prescribed prone positioning
  * Tense ascites
  * Severe abdominal pain
  * Abdominal wound or surgery
  * Pregnancy
  * Agitated delirium
* Prior intubation during hospital stay
* Cardiogenic pulmonary edema
* Exacerbation of asthma or COPD
* Chronic lung disease, including:

  * Interstitial lung disease
  * Cystic fibrosis
  * Lung mass, lung cancer, or metastasis to the lung
  * Lung transplant recipient
  * Any disease that requires home oxygen
* Glasgow coma score < 15
* Chest tube, pneumothorax, or pneumomediastinum
* Hemodynamic instability (mean arterial pressure < 55 mmHg or norepinephrine-equivalent vasopressor requirement > 0.1mcg/kg/min)
* Implantable electrical device (e.g. pacemaker, defibrillator, neurostimulator)
* Unreliable pulse-oximetry tracing
* Imminent intubation
* Anticipated lack of patient availability to complete study procedures (e.g. due to planned clinical procedure such as CT scan or dialysis during potential time of study)
* Attending physician refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in SpO2/FiO2 | At the end of each treatment period, up to 45 minutes
  The change in SpO2/FiO2 within each participant as measured at baseline and at the end of each treatment assignment period. The average SpO2/FiO2 over the last five minutes of the treatment period will be used.

SECONDARY OUTCOMES:
Change from baseline in Respiratory Rate | At the end of each treatment period, up to 45 minutes
  The change in Respiratory Rate within each participant as measured at baseline and at the end of each treatment assignment period. The average Respiratory Rate over the last five minutes of the treatment period will be used.
Change from baseline in ROX Index | At the end of each treatment period, up to 45 minutes
  The change in ROX index within each participant as measured at baseline and at the end of each treatment assignment period. ROX index is calculated as SpO2/FiO2 divided by the Respiratory Rate. The average ROX index over the last five minutes of the treatment period will be used.
Change from baseline in Transcutaneous Carbon Dioxide (CO2) | At the end of each treatment period, up to 45 minutes
  The change in Transcutaneous Carbon Dioxide within each participant as measured at baseline and at the end of each treatment assignment period. The average Transcutaneous Carbon Dioxide over the last five minutes of the treatment period will be used.
Change from baseline in Heart Rate | At the end of each treatment period, up to 45 minutes
  The change in Heart Rate within each participant as measured at baseline and at the end of each treatment assignment period. The average Heart Rate over the last five minutes of the treatment period will be used.
Change from baseline in Blood Pressure | At the end of each treatment period, up to 45 minutes
  The change in Blood Pressure within each participant as measured at baseline and at the end of each treatment assignment period. The average Blood Pressure over the last five minutes of the treatment period will be used.
Change from baseline in Breathing Discomfort | At the end of each treatment period, up to 45 minutes
  The change in Breathing Discomfort within each participant as measured at baseline and at the end of each treatment assignment period. Breathing Discomfort will be measured with component A1 of the Multidimensional Dyspnea Profile.
Change from baseline in Lightheadedness | At the end of each treatment period, up to 45 minutes
  The change in Lightheadedness within each participant as measured at baseline and at the end of each treatment assignment period. Lightheadedness will be measured with an ordinal scale ranging from 0 to 10.
Change from baseline in Nausea | At the end of each treatment period, up to 45 minutes
  The change in Nausea within each participant as measured at baseline and at the end of each treatment assignment period. Nausea will be measured with an ordinal scale ranging from 0 to 10.
Change from baseline in Skin Discomfort | At the end of each treatment period, up to 45 minutes
  The change in patient-reported Skin Discomfort as measured at baseline and at the end of each treatment assignment period. Skin Discomfort will be measured with an ordinal scale ranging from 0 to 10.
Change from baseline in Skin Erythema | At the end of each treatment period, up to 45 minutes
  The change in Skin Erythema within each participant as measured at baseline and at the end of each treatment assignment period. Skin erythema will be measured by investigator visual assessment using a five-point scale.
Tolerance of intervention period | For the duration of each treatment period, up to 45 minutes
  Patient able to complete the entire treatment period of intervention without early discontinuation for intolerance
Proportion of time within 3 cm H2O of target CNEP level | For the duration of each treatment period, up to 45 minutes
  Ability to reach and maintain the target CNEP level, defined as CNEP within ± 3 cm H2O of the prescribed value
Proportion of time within 5 cm H2O of target CNEP level | For the duration of each treatment period, up to 45 minutes
  Ability to reach and maintain the target CNEP level, defined as CNEP within ± 5 cm H2O of the prescribed value

OTHER OUTCOMES:
Change from baseline in other components of the Multidimensional Dyspnea Profile | At end of study
  The change in other components of the Multidimensional Dyspnea Profile within each participant as measured at baseline and at the end of the study. At end of study, participants will be instructed to consider their breathing on average during CNEP to obtain the post-baseline measure.
Change from baseline in Tidal Volume | At the end of each treatment period, up to 45 minutes
  The change in Tidal Volume within each participant as measured at baseline and at the end of each treatment assignment period, estimated from lung electrical impedance tomography. The average Tidal Volume over the last five minutes of the treatment period will be used.
Change from baseline in End-Expiratory Lung Volume | At the end of each treatment period, up to 45 minutes
  The change in End-Expiratory Lung Volume within each participant as estimated from end-expiratory lung impedance measured at baseline and at the end of each treatment assignment period. The average End-Expiratory Lung Impedance over the last five minutes of the treatment period will be used to derive change in end-expiratory lung volume.
Change from baseline in Minute Ventilation | At the end of each treatment period, up to 45 minutes
  The change in Minute Ventilation within each participant as measured at baseline and at the end of each treatment assignment period, estimated from lung electrical impedance tomography. The average Minute Ventilation over the last five minutes of the treatment period will be used.
Change from baseline in Anteroposterior Ventilation Ratio | At the end of each treatment period, up to 45 minutes
  The change in Anteroposterior Ventilation Ratio within each participant as measured at baseline and at the end of each treatment assignment period, estimated from lung electrical impedance tomography. The average Anteroposterior Ventilation Ratio over the last five minutes of the treatment period will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Beitler, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes